CLINICAL TRIAL: NCT03963323
Title: GLANCE2.1 - Glucosamine and Chondroitin (G&C) Effects Study
Brief Title: Glucosamine and Chondroitin in Gut in Preventing People From Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: RG1001759; 8645 (Other: FHCRC)
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Glucosamine; Chondroitin Sulfates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (glucosamine sulfate/chondroitin sulfate tablet) (Experimental): Patients receive glucosamine sulfate/chondroitin sulfate tablet PO on days 1-14 in the absence of disease progression or unacceptable toxicity. Fourteen days later, patients crossover to Arm II.
  Interventions: Dietary Supplement: Glucosamine Sulfate/Chondroitin Sulfate Tablet
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO on days 1-14 in the absence of disease progression or unacceptable toxicity. Fourteen days later, patients crossover to Arm I.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Glucosamine Sulfate/Chondroitin Sulfate Tablet — Given PO
  Arms: Arm I (glucosamine sulfate/chondroitin sulfate tablet)
Other: Placebo — Given PO
  Other Names: PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This trial studies glucosamine and chondroitin in preventing inflammation. Glucosamine and chondroitin often used as a dietary supplement to promote joint health may have a preventive role in inflammation and cancer. This trial may help identify the bacteria that help process them in the gut.

ELIGIBILITY:
Inclusion Criteria:

- From the Greater Seattle area

Exclusion Criteria:

* Chronic medical illness, history of gastrointestinal, hepatic, or renal disorders, or inflammatory conditions (including autoimmune and inflammatory diseases)
* Pregnancy or lactation
* Currently on a weight-loss diet
* Alcohol intake of greater than 2 drinks/day (2 drinks being equivalent to 720 ml beer, 240 ml wine or 90 ml spirits)
* Current use of prescription or over-the-counter medications other than oral contraceptives and hormone secreting intrauterine device (IUD)s, multivitamin pills or infrequent use of aspirin and nonsteroidal anti-inflammatory drugs (NSAIDs), or use of aspirin or NSAIDs more than 2 days per week
* Abnormal renal, liver or metabolic test
* Inability to swallow pills
* Known allergy to shellfish
* Not willing to take pills made from shellfish or animal sources
* Intention to relocate out of study area within next 2 months
* Any antibiotic use in the past 6 months

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants that experienced a shift in bacterial community assessed by operational taxonomic units | Up to 2 years
  Shifts in the bacterial communities is based on clustering of operational taxonomic units (OTU) at 97% similarity

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Lampe, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No